CLINICAL TRIAL: NCT01211574
Title: Pilot Study Testing Professional, Peer, and Mentor Health Coaches for Weight Loss
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Tricia M. Leahey, Ph.D., Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2044-10
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (3):
- peer coach (Experimental): Participants will be coached by a peer between treatment visits.
  Interventions: Behavioral: peer coach
- mentor (Experimental): Participants will be coached by a mentor between treatment visits
  Interventions: Behavioral: mentor
- Professional (Experimental): Participants will be coached by an interventionist between treatment visits
  Interventions: Behavioral: Professional

INTERVENTIONS:
Behavioral: peer coach — Participants will receive behavioral weight loss treatment and be coached by a peer between treatment visits.
  Arms: peer coach
Behavioral: mentor — Participants will receive behavioral weight loss treatment and be coached by a mentor between treatment visits.
  Arms: mentor
Behavioral: Professional — Participants will receive behavioral weight loss treatment and be coached by a behavioral weight loss interventionist between treatment visits.
  Arms: Professional

SUMMARY:
Participants will be randomly assigned to 1 of 3 types of health coaches, Peers, Mentors, or Professionals. The aim of this study is to examine the feasibility and preliminary efficacy of health coaching for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* age 40-60

Exclusion Criteria:

* Participants will be excluded if they:

  1. Are unwilling to participate in a weight control program that includes weight coaches.
  2. Report not being able to walk 2 blocks (1/4 mile) without stopping.
  3. Are participating in a weight loss program, taking a weight loss medication, have a history of bariatric surgery, or lost ≥ 5% of body weight during the past 6-months.
  4. Are pregnant, lactating, less than 6 months post-partum or plan to become pregnant during the time of the intervention.
  5. Report a heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Participants reporting joint problems, medication use, or other medical conditions that may limit their ability to exercise will be required to obtain written permission from their physician to participate in the intervention.
  6. Report conditions that, in the judgment of the PI, would render the participant unlikely to follow the study protocol (e.g., terminal illness, relocation, substance abuse, bulimia nervosa, dementia, or severe psychiatric condition).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
weight change | 0 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tricia M Leahey, PhD, Principal Investigator — The Miriam Hospital / Warren Alpert Medical School at Brown University